CLINICAL TRIAL: NCT05471258
Title: Efficacy of Therapy Using Monopolar Dielectric by Radiofrequency on the Symptoms of Myofascial Trigger Points in Patients With Chronic Non-specific Low Back Pain.
Brief Title: Efficacy of Therapy Using Monopolar Dielectric Radiofrequency Signals on the Symptoms of Myofascial Trigger Points in Patients With Chronic Nonspecific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UALBIO2021/005
Record Dates: First submitted 2022-03-14; First posted 2022-07-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
Keywords: chronic low back pain; monopolar dielectric diathermy; placebo; randomised double-blind clinical trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Once the study is over, the control group will have the opportunity to receive radiofrequency treatment for three weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not familiar with diathermy, and will lie prone while receiving treatment. They will also be cited on different days of the week to the experimental group.
  The therapist assessing the outcome measures does not know which group the patients belong to, and will be supervised by the principal investigator so that they do not ask any questions about it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: monopolar dielectric diathermy (Experimental): The Experimental Group formed by 30 subjects will undergo an application of monopolar electrical diathermy by radiofrequency emission (MDR) using the Physicalm® device developed by the electro-medicine company Biotronic Advance Develops SL, on the lumbar muscles by means of rotary movements and translation, adapting to the muscle fibers of the lumbar area. A pulsed emission of 840 KHz and 30v will be made dynamically during a treatment time of 20 minutes. 3 weekly sessions will be performed for 3 weeks, a total of 9 treatment sessions.
  Interventions: Other: Experimental: monopolar dielectric diathermy
- Placebo (Placebo Comparator): The 30 participants in the control group will receive a placebo treatment, consisting of the same execution protocol as the EG, but with a non-emitting device whose software and hardware will be exactly the same as that used in the EG. The intervention will be simulated for 20 minutes.
  3 weekly sessions will be held for 3 weeks, a total of 9 treatment sessions.
  Interventions: Other: Control: Placebo

INTERVENTIONS:
Other: Experimental: monopolar dielectric diathermy — The Experimental Group formed by 30 subjects will undergo an application of monopolar electrical diathermy by radiofrequency emission (MDR) using the Physicalm® device developed by the electro-medicine company Biotronic Advance Develops SL, on the lumbar muscles by means of rotary movements and translation, adapting to the muscle fibers of the lumbar area. A pulsed emission of 840 KHz and 30v will be made dynamically during a treatment time of 20 minutes. 3 weekly sessions will be performed for 3 weeks, a total of 9 treatment sessions.
  Arms: Experimental: monopolar dielectric diathermy
Other: Control: Placebo — The 30 participants in the control group will receive a placebo treatment, consisting of the same execution protocol as the EG, but with a non-emitting device whose software and hardware will be exactly the same as that used in the EG. The intervention will be simulated for 20 minutes.
  3 weekly sessions will be held for 3 weeks, a total of 9 treatment sessions.
  Arms: Placebo

SUMMARY:
A total of 74 people diagnosed with non-specific chronic low back pain of more than 3 months of evolution and who are not currently undergoing any type of treatment will be recruited, with ages between 35 and 65 years. A random distribution will be made into two treatment groups (monopolar diathermy by radiofrequency versus placebo). Participants will receive treatment three per week for a period of three weeks, in the physiotherapy laboratories of the University of Almería, with a follow-up evaluation post-intervention (one months) and two months after the end of treatment. At their first visit, participants will be screened for study eligibility according to the study inclusion and exclusion criteria, and will be evaluated by a therapist blinded to the intervention. After this face-to-face evaluation, patients will be randomly assigned to one of the two groups and will receive treatment for low back pain according to their random assignment group by two therapists belonging to the research group and trained in the techniques used.

DETAILED DESCRIPTION:
The technique of applying monopolar electrical diathermy by radiofrequency emission (MDR), using the Physicalm® device, allows electromagnetic waves to be applied transcutaneously in a capacitive and monopolar manner, making focused energy deposits in the areas compromised with the painful process. The intervention with this device consists of different independent programs adapted to the different modalities of clinical pain. Through adaptations of the digitally modulated electromagnetic signals in terms of their intensity, frequency, form and duration, analgesia and pain relief can be obtained in different conditions musculoskeletal.

Despite being a clinical electrotherapy technique currently widely used by physiotherapists, there are few clinical trials on the application of monopolar electrical diathermy by radiofrequency emission (MDR) in ailments of lumbar origin caused by myofascial trigger points. The difference with other systems that use high-frequency electrophysical agents such as short waves or microwaves lies mainly in the ability to penetrate the tissues, producing a thermal effect at a greater depth.

Due to all the structural and functional alterations that occur in chronic non-specific low back pain, this randomized clinical trial project was born, with the aim of providing an answer to the disabling symptoms suffered by patients with chronic non-specific low back pain, searching for tools of safe and effective treatment from the field of Physiotherapy, which report a benefit in the symptoms, functionality and quality of life of patients diagnosed with chronic non-specific low back pain caused by PGM.

A total of 74 people diagnosed with non-specific chronic low back pain of more than 3 months of evolution and who are not currently undergoing any type of treatment will be recruited, with ages between 35 and 65 years. A random distribution will be made into two treatment groups (monopolar diathermy by radiofrequency versus placebo).

The 37 subjects of the experimental group (EG) will receive an application of monopolar electrical diathermy by radiofrequency emission (MDR) by means of the Physicalm® device (developed by the electro-medicine company Biotronic Advance Develops SL), on the lumbar muscles by means of rotary movements and translation, adapting to the muscle fibers of the lower back, contacting and applying the treatment to the active myofascial trigger points of the following muscles: quadratus lumborum, multifidus and iliocostalis, following the PGM maps described by Travell and Simons. A pulsed emission of 840 KHz and 30v will be carried out dynamically for a treatment time of 20 minutes. 3 weekly sessions will be performed for 3 weeks, a total of 9 treatment sessions.

The 37 subjects in the control group (CG) will be administered a placebo treatment consisting of the same execution protocol as the EG, but with a non-emitting device whose software and hardware will be exactly the same as that used in the EG. The intervention will be simulated for 20 minutes.

A pulsed emission of 840 KHz and 30v will be carried out dynamically for a treatment time of 20 minutes. 3 weekly sessions will be performed for 3 weeks, a total of 9 treatment sessions.

The outcome assessor and study statistician will be blinded throughout the entire process.

A baseline assessment of the primary and secondary outcome measures will be performed before randomization of the participants to the different groups, an immediate post-treatment assessment (1 day after the last intervention) and an assessment two months after the end of the procedure intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* LBP for/over three months
* Age between 30 and 65 years
* Score equal or superior of four points on the Roland Morris Disability
* Questionnaire Not currently receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis;
* Any clinical signs of radiculopathy;
* Diagnosis of spondylolisthesis;
* Diagnosis of fibromyalgia;
* Treatment with corticosteroid or oral medication within the past two weeks;
* A history of spinal surgery;
* Contraindication for MDR;
* Disease of the central or peripheral nervous system; (9) Patients with cardiac complications and / or patients who have recently undergone radiotherapy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in pressure algometry (Wagner Algometer) in myofascial trigger points assessment of pressure pain threshold. | At baseline, at 4 weeks and at 2 months
  The algometer consists of a rubber tip and a dial that measures the pressure applied to the MTrP in increments of 0.5 kg. Three measurements were performed for each one of the selected trigger points: iliocostal muscle level L1; multifidus level L2, S1 and S4; quadratus lumbar PGM deep superior, deep inferior, superficial superior and superficial inferior. The average value of 3 repetitive measurements with intervals of 30 to 60 seconds was used for statistical analysis.
Change from baseline in pain intensity. Visual analogue scale. | At baseline, at 4 weeks and at 2 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain
Change from baseline in Roland Morris Disability Questionnaire (RMDQ). | At baseline, at 4 weeks and at 2 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 4 weeks and at 2 months
  It has 10 items associated to activities of daily living, each ítem has a puntuation fron 0 to 5 points.
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, at 4 weeks and at 2 months
  Is a 17-item questionnaire that measures the fear of movement and (re)injury. Ratings are summed to yield a total score (ranging from 17-68 points) where higher values reflect greater fear of (re)injury.
Change from baseline on Quality of Life. SF-36 Health questionnaire | At baseline, at 4 weeks and at 2 months
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test. | At baseline, at 4 weeks and at 2 months
  It measures the isometric endurance of trunk flexion muscles.
Change from baseline in lumbar mobility flexion | At baseline, at 4 weeks and at 2 months
  For the quantification of lumbar flexion an angular inclinometer is used (Fleximeter UM 8320-3 RJ Code Research Institute, Brazil).
Change from baseline of Pittsburgh Sleep Quality Index (PSQI) | At baseline, at 4 weeks and at 2 months
  Is a 10-item questionnaire with a total of 19 questions related to sleep habits in the previous month. The questions are divided into 7 areas, each with a score of between 0 and 3 points.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro Sánchez, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- Adelaida María Castro Sánchez, Almería, Almeria, Spain

REFERENCES:
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Adamson J, Hunt K, Nazareth I. The influence of socio-demographic characteristics on consultation for back pain--a review of the literature. Fam Pract. 2011 Apr;28(2):163-71. doi: 10.1093/fampra/cmq085. Epub 2010 Oct 25. PMID 20974654
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Kumaran B, Watson T. Thermal build-up, decay and retention responses to local therapeutic application of 448 kHz capacitive resistive monopolar radiofrequency: A prospective randomised crossover study in healthy adults. Int J Hyperthermia. 2015;31(8):883-95. doi: 10.3109/02656736.2015.1092172. Epub 2015 Nov 2. PMID 26524223
- [Background] Úbeda A, Hernández-Bule ML, Trillo MA, Cid MA, Leal J. Cellular response tonon-thermal doses of radiofrequency currents used in electro-thermaltherapy. J Jpn Soc Laser Surg Med. 2006;27(3):187.31.
- [Background] Tashiro Y, Hasegawa S, Yokota Y, Nishiguchi S, Fukutani N, Shirooka H, Tasaka S, Matsushita T, Matsubara K, Nakayama Y, Sonoda T, Tsuboyama T, Aoyama T. Effect of Capacitive and Resistive electric transfer on haemoglobin saturation and tissue temperature. Int J Hyperthermia. 2017 Sep;33(6):696-702. doi: 10.1080/02656736.2017.1289252. Epub 2017 Feb 19. PMID 28139939
- [Background] Kumaran B, Watson T. Radiofrequency-based treatment in therapy- related clinical practice - a narrative review. Part II: chronic conditions. Phys Ther Rev. 2016;20:325-343
- [Background] Albornoz-Cabello M, Barrios-Quinta CJ, Escobio-Prieto I, Sobrino-Sanchez R, Ibanez-Vera AJ, Espejo-Antunez L. Treatment of Patellofemoral Pain Syndrome with Dielectric Radiofrequency Diathermy: A Preliminary Single-Group Study with Six-Month Follow-Up. Medicina (Kaunas). 2021 Apr 28;57(5):429. doi: 10.3390/medicina57050429. PMID 33925211
- [Background] Ibanez-Vera AJ, Garcia-Romero JC, Alvero-Cruz JR, Lomas-Vega R. Effects of Monopolar Dielectric Radiofrequency Signals on the Symptoms of Fibromyalgia: A Single-Blind Randomized Controlled Trial. Int J Environ Res Public Health. 2020 Apr 3;17(7):2465. doi: 10.3390/ijerph17072465. PMID 32260313
- [Result] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712